CLINICAL TRIAL: NCT00288327
Title: Testing Lifestyle Interventions for CVD Risk Reduction in Older, Underserved Women; Enhanced WISEWOMAN Project
Brief Title: NC Enhanced WISEWOMAN Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); North Carolina Department of Health and Human Services (Other Government)
Responsible Party: Alice Ammerman, DrPH, RD/Director, Center for Health Promotion and Disease Prevention
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: U48/CCU409660
Record Dates: First submitted 2006-02-06; First posted 2006-02-07 (Estimated); Last update posted 2009-03-13 (Estimated); Status verified 2009-03

CONDITIONS: Cardiovascular Disease
Keywords: diet; physical activity; smoking cessation
MeSH Terms: conditions — Cardiovascular Diseases; Motor Activity; Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Enhanced New Leaf Intervention
  Interventions: Behavioral: Lifestyle behavior change program
- 2 (Other): Minimum Intervention
  Interventions: Behavioral: Pamphlets

INTERVENTIONS:
Behavioral: Lifestyle behavior change program — Intervention included a six-month intensive intervention of 2 individual counseling sessions, 3 group sessions, and 3 phone calls from a peer counselor followed by a maintenance phase (6 months) including 1 individual counseling session and 7 monthly peer counselor calls.
  Arms: 1
Behavioral: Pamphlets — Nutritional and physical activity pamphlets from American Heart Association
  Arms: 2

SUMMARY:
The overall aim of the study was to test the feasibility and effectiveness of a cardiovascular disease risk reduction intervention program for midlife, low-income women. We enhanced an existing nutrition and physical activity intervention tool, A New Leaf...Choices for Healthy Living, which was designed specifically for this demographic group as part of the CDC's WISEWOMAN Program. The enhanced intervention was tested in a randomized controlled trial in a community health center setting.

DETAILED DESCRIPTION:
We conducted a 2 year study to test the feasibility and effectiveness of a CVD risk reduction intervention program for older, under or uninsured women. We used an existing nutrition and physical activity (PA) intervention tool (New Leaf…Choices for Healthy Living) designed specifically for this demographic group as part of the WISEWOMAN program (A CDC-funded CVD risk factor screening and intervention program for older, low-income women). We enhanced this already tested intervention to include: 1) the latest recommendations regarding dietary fat and carbohydrate intake, 2) group education sessions and follow-up telephone contacts from lay health advisors (LHAs); and 3) a community resource linkage component delivered primarily by LHAs. We tested the enhanced intervention in a randomized controlled trial in a community health center setting.

A total of 240 women aged 40-64 were randomized to the enhanced New Leaf intervention or minimum intervention groups. Women in the enhanced New Leaf group received a 6 month intensive intervention consisting of 2 individual counseling sessions at the CHC, postcard mailings, 3 group sessions, and lay health advisor (LHA) guided linkages to community resources for diet and PA. This was followed by a 6 month maintenance period led by the LHA and including 6 phone contacts, and 3 tailored mailings along with continued community resource linkages. Primary outcome measures at 6 and 12 months included 1) PA measured by CSA accelerometer and 2) fruit, vegetable, and fat intake. Secondary outcomes included biomarkers of dietary intake (red blood cell membrane fatty acids, carotenoids), CVD risk factors (total and HDL cholesterol, blood pressure), and psychosocial variables.

ELIGIBILITY:
Inclusion Criteria:

* Women 40-64 years old
* Patient at participating site who is considered an appropriate candidate by the primary care clinician
* Ability and willingness to provide informed consent
* Availability for follow-up--plan to reside within 50 miles of study site for 1 year
* Home phone or easy access to phone

Exclusion Criteria:

* Medical condition for which intervention may not be appropriate
* Pregnancy/lactation
* Severe chronic medical conditions such that interventions to improve diet and physical activity are not appropriate

Ages: 40 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 258 (Actual)
Dates: Start 2003-03; Primary Completion 2004-12 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
physical activity
fruit intake
vegetable intake
fat intake

SECONDARY OUTCOMES:
Biomarkers of dietary intake (red blood cell membrane fatty acids, carotenoids);
CVD risk factors (total and HDL cholesterol, blood pressure);
Psychosocial variables

CONTACTS AND LOCATIONS:
Overall Officials: Alice S Ammerman, DrPH, RD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- New Hanover Community Health Center, Wilmington, North Carolina, United States

REFERENCES:
- [Background] Rosamond WD, Ammerman AS, Holliday JL, Tawney KW, Hunt KJ, Keyserling TC, Will JC, Mokdad AH. Cardiovascular disease risk factor intervention in low-income women: the North Carolina WISEWOMAN project. Prev Med. 2000 Oct;31(4):370-9. doi: 10.1006/pmed.2000.0726. PMID 11006062
- [Derived] Keyserling TC, Samuel Hodge CD, Jilcott SB, Johnston LF, Garcia BA, Gizlice Z, Gross MD, Savinon CE, Bangdiwala SI, Will JC, Farris RP, Trost S, Ammerman AS. Randomized trial of a clinic-based, community-supported, lifestyle intervention to improve physical activity and diet: the North Carolina enhanced WISEWOMAN project. Prev Med. 2008 Jun;46(6):499-510. doi: 10.1016/j.ypmed.2008.02.011. Epub 2008 Feb 15. PMID 18394692